CLINICAL TRIAL: NCT05092776
Title: International, Multicenter, Double Blind, Placebo-controlled, Randomized Clinical Study of Efficacy and Safety of RPH-104 for Resolution and Prevention of Recurring Attacks in Adult Subjects With Familial Mediterranean Fever With Resistance to or Intolerance of Colchicine
Brief Title: Efficacy and Safety of RPH-104 for Resolution and Prevention of Recurring Attacks in Adult Subjects With Familial Mediterranean Fever With Resistance to or Intolerance of Colchicine
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: Data Management 365 (Industry); Atlant Clinical LLC (Unknown); R-Pharm JSC (Unknown); Unimed Laboratories (Industry); Exacte Labs LLC (Industry); Key Stat LLC (Unknown); TRPharm İlaç Sanayi Ticaret Anonim Şirketi and ASCOT SCIENCE Education and Consulting Ltd. (Unknown); Ascot Eğitim ve Danışmanlık LTD. ŞTİ. (Unknown)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL04018065
Record Dates: First submitted 2021-09-09; First posted 2021-10-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Familial Mediterranean Fever; FMF
Keywords: RPH-104; colchicine inefficacy; colchicine intolerance; subcutaneous
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPH-104 (Experimental): Test product group receiving RPH-104 subcutaneous (s.c.) injections:160 mg on Day 0, 80 mg on Day 7, Day 14 and every 2 weeks (q2w) thereafter.
  In case "marker" attack does not resolve at Visit 2 - the treatment group will be unblinded: patients will receive planned RPH-104 80 mg administration.
  In case of a new attack on further days of treatment period until Visit 10 inclusive - the treatment group will be unblinded: the dose of RPH-104 could be escalated to 160 mg q2w; The patients already receiving RPH-104 160 mg q2w will continue to receive RPH-104 at this dose. Further dose escalation is forbidden.
  Interventions: Biological: RPH-104
- Placebo (Placebo Comparator): Placebo group receiving the equivalent placebo dose also as s.c. injections on Day 0, Day 7, Day 14 and q2w thereafter.
  In case the "marker" attack does not resolve at Visit 2 - the treatment group will be unblinded: patients will be switched to active treatment with RPH-104 in SC injections at a dose of 160 mg followed by administration of 80 mg in 7 days at the Attack + 7 days Visit, and 80 mg at the next Visits.
  In a case of a new attack the patients switching from placebo and receiving RPH-104 at 80 mg dose could be escalated to RPH-104 160 mg q2w; Further dose escalation is forbidden.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RPH-104 — solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL glass vial
  Arms: RPH-104
Drug: Placebo — Normal Saline (0.9% Sodium Chloride solution for subcutaneous Injection), 2 mL in the 4 mL-glass vial. The placebo will contain no active pharmaceutical ingredients.
  Arms: Placebo

SUMMARY:
Study purpose is an evaluation of efficacy and safety of RPH-104 in the population of subjects with Familial Mediterranean Fever (FMF) with colchicine resistance or intolerance(i.e. colchicine resistant (crFMF).. Primary objective is to determine proportion of subjects with complete response to treatment with RPH-104 compared to placebo among FMF subjects with colchicine resistance or intolerance.

DETAILED DESCRIPTION:
The study is supposed to enroll (randomize) (n= not less than 28, not less than 14 per group), so that not less than 24 to complete study in full (including all the treatment period visits and follow-up period visits - Visit 11 for patients who agreed to participate in the Open-label extension (OLE) study; Visit 11 and Visit 12 for those who do not wish to participate in the OLE study; given potential withdrawal at screening the number of screened subjects (signed Informed Consent Form (ICF) is planned to be up to 84.

The study will consists of three following periods:

1. Screening period (up to 12 weeks); Throughout the screening the subjects will be monitored to identify "marker" attacks and verify the subject eligibility. The subjects having an attack during screening period and meeting inclusion/exclusion criteria will be enrolled into treatment period.
2. Double-blind randomized placebo-controlled treatment period (16 weeks);

   The subjects enrolled will be randomized to one of the treatment groups in 1:1 ratio:
   * RPH-104 group to receive subcutaneous (SC) injections according to the following regimen: 160 mg on Day 0, 80 mg on Day 7, Day 14 and once every 2 weeks (q2w) thereafter;
   * placebo group to receive matching SC injections on Day 0, Day 7, Day 14 and q2w thereafter.

   Efficacy assessment will be performed at Visit 2 and Visit 3, and subsequently every 2 weeks up to Visit 10 inclusive; safety assessment will be performed throughout the study (Visit 1 - Visit 12). In a case of adverse event (AE) development (or other safety reasons), additional unscheduled safety visits could be performed throughout the study. Starting from Visit 2, additional unscheduled visits due to suspected development of FMF attack could be performed. In a case of a recurrent attack, the patient should come to the study site within 2 days from the attack onset for the attack registration.

   The treatment response (i.e. the resolution of FMF "marker" attack/absence of recurrent attacks) will be assessed throughout the treatment period with the investigational products administered both blind and open-label. Responders will continue the study treatment with the assigned investigational products (RPH-104 or placebo as a single SC 2 mL injection q2w, based on the randomization group) in a blinded manner. In non-responders, the following treatment modifications are possible:
   * In a case the "marker" attack has not resolved by Visit 2 - the treatment group will be unblinded:

     * patients from placebo group will be switched to active treatment with RPH-104 in SC injections at a dose of 160 mg (single dose, first injection) followed by administration of 80 mg in 7 days at the Attack + 7 days Visit (with procedures corresponding to Visit 2), and 80 mg at the next scheduled Visit performed 1 week later than initially scheduled (with procedures corresponding to this Visit) after the Attack + 7 days Visit.
     * patients from RPH-104 group will receive planned RPH-104 80 mg administration.
   * In a case of recurrent FMF attack confirmation at a scheduled visit - the treatment group will be unblinded (if still blinded):

     * patients from placebo group will be switched to active treatment with RPH-104 in SC injections at a dose of 160 mg (single dose, first injection) followed by administration of 80 mg in 7 days at the Attack + 7 days Visit (with procedures corresponding to Visit 2), and then at the next scheduled Visit (with procedures corresponding to the further study schedule) and all the next scheduled visits every 2 weeks thereafter;
     * patients from RPH-104 group or patients who were switched from placebo group and receiving RPH-104 80 mg will receive RPH-104 160 mg administration at the visit and thereafter 160 mg q2w;
     * patients already receiving RPH-104 160 mg q2w in unblinded manner can continue treatment or can discontinue treatment at the discretion of Investigator, based on the risk/benefit assessment of the further RPH-104 treatment.
   * In a case of recurrent FMF attack confirmation at an unscheduled visit - the treatment group will be unblinded (if still blinded):

     * if a recurrent FMF attack is recorded and the subject visits the study site within 3 days before the next scheduled visit (starting from Visit 3), the subject will undergo all the next scheduled visit procedures including the unblinded RPH-104 administration and blood sampling provided for at this scheduled visit. The treatment rules for a scheduled visit described above are applicable in this case;
     * in a case of a recurrent attack and subject's arrival to the site more than 3 days before the next scheduled visit but not less than 7 days after the previous scheduled visit (starting from Visit 2), the unscheduled visit will be performed on the day of arrival to the study site (and the administration will be shifted from the planned next scheduled visit). The treatment rules for a scheduled visit described above are applicable in this case. Further the subject will not attend the next scheduled visit and all the visit procedures per Protocol should be performed as an unscheduled visit. Afterwards, the initially planned visits schedule for a patient will be kept;
     * in a case of unscheduled visit within 7 days after administration of the scheduled blinded RPH-104 80 mg dose or placebo all procedures planned for unscheduled visit to be performed. If at such unscheduled visit development of a recurrent attack is confirmed the subject will be unblinded:

       * patients from placebo group will be switched to active treatment with RPH-104 in SC injections at the unscheduled visit at a dose of 160 mg (single dose, first injection) followed by administration of 80 mg in 7 days at the Attack + 7 days Visit (with procedures corresponding to Visit 2), and 80 mg at the next scheduled Visit performed 1 week later (with procedures corresponding to this Visit) after the Attack + 7 days Visit;
       * patients from RPH-104 group or patients who were switched from placebo group and receiving RPH-104 80 mg q2w will receive RPH-104 80 mg administration at the visit and thereafter 160 mg q2w starting from the next scheduled visit;
       * patients already receiving RPH-104 160 mg q2w will not receive RPH-104 at this unscheduled visit and can continue treatment or can discontinue treatment at the discretion of Investigator, based on the risk/benefit assessment of the further RPH-104 treatment.

   For patients receiving RPH-104 at a dose of 160 mg q2w no further dose escalation is carried out. In a case of consequent recurrent attacks this patient may continue treatment with RPH-104 at a maximum dose of 160 mg q2w according to the Investigator's reasonable decision until the end of the study treatment period. No dose reduction of the investigational products could be made throughout the study.

   Maximum treatment duration is 16 weeks.

   Subjects receiving both blinded and unblinded therapy will undergo regular evaluation of efficacy and safety; the visits will be performed every 2 weeks for this purpose.

   At the last visit of the treatment period (Visit 10) after completion of all visit procedures the patients will be invited to proceed in a long-term open-label extension (OLE) study to evaluate the safety and efficacy study of RPH-104 (CL04018071).
3. Follow-up period (8 weeks) that includes safety monitoring for 8 weeks after the last dosing with the investigational products.

In case of lacking relevant clinical response and if the subjects do not wish to participate in the open-label study, they should complete all safety follow-up visits.

Therefore, the total maximum duration of participation of one patient in the study will be 37 weeks, id est (i.e.) about 9 months (1 additional week could be added to the overall study duration in case of switching from the placebo to the RPH-104 treatment for a subject due to the disease attack).

ELIGIBILITY:
Inclusion criteria:

* Presence of voluntarily signed and dated ICF to participate in this study.
* Verified diagnosis of familial Mediterranean fever (FMF) based on Tel HaShomer diagnostic criteria (Pras M., 1998) or the criteria developed by the Eurofever /Pediatric Rheumatology International Trials Organization (PRINTO) expert group (2019);
* Presence of at least one mutation in Mediterranean fever gene (MEFV) exon 10 (results of the study performed earlier at any time may be provided or a respective test should be performed during the screening);
* Presence (at screening onset) of data on history of at least one (on average) disease attack per month throughout the last 3 months (Ozen et al., 2020);
* Presence of at least one of the below-mentioned (at screening onset) documented data confirming:

  * resistance to colchicine at the maximum tolerable therapeutic dose (up to 3 mg/day) confirmed by at least one monthly attack (on average) despite the therapy specified within at least 3 last months. Colchicine administration will be continued at stable dose if it is not associated with unacceptable adverse reactions;
  * intolerance of therapeutic or subtherapeutic doses of colchicine (unacceptable adverse reactions); Colchicine dose should be stable for at least 5 days before patient enrollment into the study (prior to screening onset).
* Ability and willingness of the subject, according to the reasonable Investigator's judgment, to attend the study site at all scheduled visits, undergo the study procedures and follow the Protocol requirements including subcutaneous (SC) injections by qualified site personnel;
* Consent of female subjects of childbearing potential defined as all females with physiological potential to conceive (except for those with absolute termination of menses to be determined retrospectively after 12 months of natural amenorrhea, i.e. amenorrhea with relevant clinical status, e.g. appropriate age) to use highly effective contraception throughout the study starting from the screening (signed ICF) and for at least 8 weeks after the study treatment completion (discontinuation); and negative pregnancy test (serum test for human chorionic gonadotropin (HCG)).

or Consent of the sexually active men subjects to use highly effective contraception throughout the study starting from the screening (signed ICF) and for at least 8 weeks after the study treatment completion (discontinuation).

A highly effective method of contraception is defined as follows:

* complete abstinence: if it corresponds to the preferred and conventional lifestyle of the female subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, postovulation method) and interrupted coitus are not considered acceptable contraceptive methods;
* female sterilization: surgical bilateral ovariectomy (with/without hysterectomy) or tubal ligation at least 6 weeks prior to the study treatment initiation. In case of ovariectomy only the female reproductive status should be verified by further hormonal test;
* male sterilization (with documented absence of sperm in ejaculate post vasectomy) at least 6 months for screening. Vasectomized male partner should be the only partner of the participating female subject;
* combination of two of the following methods (a+b or a+c or b+c):

  а) oral, injection or implanted hormonal contraceptives; in case of oral contraceptives the female subjects should administer the same product for at least 3 months prior to the study treatment;

  b) intrauterine device or contraceptive system;

  с) barrier methods: condom or occlusive cap (diaphragm or cervical cap / vaginal fornix cap) with spermicidal foam/gel/film/cream/vaginal suppository.
  * Presence of active FMF attack at Visit 1 (Day 0) lasting for not more than 2 days before Visit 1 defined as simultaneous development of clinical and serological signs of the attack including:
* Physician Global Assessment (PGA) score ≥ 2 supposing mild, moderate or severe activity of the disease (i.e. clinical signs), and
* CRP level > 10 mg/L (i.e. serological signs).

Exclusion criteria:

* Hypersensitivity to the study product (RPH-104) and/or its components/excipients.
* Administration of live (attenuated) vaccines less than 3 months prior to Day 0 (treatment initiation) and/or necessity to use such vaccine within 3 months after the study product RPH-104 treatment completion (discontinuation). Live attenuated vaccines include viral vaccines against: measles, rubella, parotitis, varicella, rotavirus, influenza (as nasal spray), yellow fever, poliomyelitis (oral polio-vaccine); tuberculosis vaccine (BCG), typhoid (oral typhoid fever vaccine) and camp fever (epidemic typhoid vaccine). Immunocompetent family members should refuse to use oral polio-vaccine throughout the subject's participation in the study.
* Conditions or signs which, according to the investigator, evidence impaired (reduced) immune response and/or significantly increase the risk of immunomodulating therapy including (but not limited to):

  * active bacterial, fungal, viral or protozoal infection at screening onset;
  * opportunistic infections and/or Kaposi's sarcoma at the screening period onset;
  * chronic bacterial, fungal or viral infection requiring systemic therapy with parenteral products at the main screening period onset;
  * human immunodeficiency (HIV), hepatitis B (HBV) or C (HCV) viral infections;
* Active tuberculosis (TB) in the history or risk factors or signs evidencing active or latent infection with M. Tuberculosis including (not limited to) the following:

  * living in specific conditions increasing the risk of contact with tuberculosis such as detention facilities, in crowded areas of person of no fixed abode, etc. within the last year before the main treatment period;
  * working in a medical institution with unprotected contact with subjects under high risk of tuberculosis or subjects with tuberculosis within the last year until the main therapy period;
  * close contact, i.e. confinement to a place (home or another confined area) for a long period of time (several days or weeks, not minutes or hours) with a subject with active pulmonary tuberculosis within the last year until the main therapy period;
  * results of examinations indicating active or latent infection with M. Tuberculosis: positive QuantiFERON-TB / T-Spot TB test at screening; chest X-ray/chest CT findings confirming pulmonary tuberculosis during screening.
* Any other relevant concomitant diseases (cardiovascular, nervous, endocrine, urinary, gastrointestinal, hepatic disorders, coagulation disorders, other autoimmune diseases, etc.) or conditions which, according to the investigator's judgment, may affect the subject's participation or well-being in the study and/or distort assessment of the study results.
* History of organ transplantation or necessity in transplantation at the screening onset.
* Any malignancies during the screening period or for 5 years before screening except for non-metastatic basal cell and squamous cell skin cancer after total resection or in situ carcinoma of any type after total resection.
* Pregnancy or breastfeeding.
* History of alcohol or psychoactive substance abuse according to the investigator's evaluation.
* Severe renal failure: creatinine clearance (ClCr) calculated using Cockcroft-Gault formula < 30 mL/min.
* Prior therapy with:

  * rilonacept - less than 6 weeks prior to Day 0 of the study;
  * canakinumab - less than 12 weeks prior to Day 0 of the study;
  * anakinra - less than 72 hours prior to Day 0 of the study;
  * rituximab - less than 24 weeks prior to Day 0;
  * tumor necrosis factor alpha (TNF-α), interleukin (IL)-6 inhibitors and other biologics - less than 6 weeks or 5 half-life periods (whichever is longer) prior to Day 0 of the study;
  * immunosuppressive drugs (azathioprine, leflunomide, dapsone, cyclosporine, mycophenolate mofetil, tacrolimus, sirolimus, mercaptopurine methotrexate, etc.) - less than 4 weeks or 5 half-lives (whichever is longer) prior to Day 0 of the study. In the case of administration of leflunomide, the completion of a course of elimination with cholestyramine should be documented;
  * intravenous (IV) immunoglobulin (Ig) - less than 8 weeks prior to Day 0;
  * use of any other biologic less than 5 half-life periods prior to Day 0 of the study;
  * IV administration of glucocorticoids less than 1 week (since the end of treatment) prior to Day 0 of the study;
  * intramuscular, intra-articular or peri-articular administration of glucocorticoids less than 4 weeks prior to Day 0;
  * systemic therapy with oral glucocorticoids at doses > 0,2 mg/kg/day equivalent to the prednisolone dose on Day 0;
  * changes in the glucocorticoids dose/dosage regimen within at least 4 weeks prior to screening.
* Any of the deviations in the laboratory tests below:

  * absolute neutrophil count < 1.5 x 10^9/L (1500 /mm^3),
  * White blood cell (WBC) count < 3 x 10^9/L (<3000/mm^3),
  * platelet count < 100 ^9/L (<100000/mm^3 or <100000×10^6/L),
  * alanine aminotransferase (ALT) and/or aspartate transaminase (AST) ≥ 2 x upper limits of normal (ULN) if at the screening ALT, AST ≥ 2 x ULN but < 3 ULN, retest is allowed,
  * bilirubin > 1.5 x ULN (except for documented cases of Gilberts syndrome).
* Parallel participation in other clinical studies at the screening onset or administration of any unauthorized (investigational) products less than 4 weeks or 5 half-life periods (whichever is longer) before Visit 1 (treatment initiation).
* Previous participation in this clinical study, in case of passing the randomization procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with complete response during 16 week therapy with RPH-104 vs. placebo in FMF subjects with colchicine inefficacy or intolerance. | Up to 16 weeks
  Complete response defined as resolution of "marker" attack by Visit 2 (Day 7) and lack of recurrent attacks during the treatment period up to Visit 10 (Day 112).
  Criteria of resolution of a "marker" FMF attack include simultaneous clinical and laboratory signs of the attack resolution:
  * Physician Global Assessment (PGA) score < 2 (i.e. minimum or complete lack of clinical signs and symptoms) AND
  * C-reactive protein (CRP) level ≤ 10 mg/L OR CRP reduction by ≥ 70% compared to baseline defined at enrollment to treatment period (Visit 1).
  Criteria of a recurrent FMF attack development after resolution of "marker" attack include simultaneous development of clinical and laboratory signs of the attack:
  * PGA score ≥ 2 assuming mild, moderate or severe disease activity (i.e. clinical signs), AND
  * CRP level ≥ 30 mg/L (serological signs).
  PGA is a 5-point scale: from 0 = no disease-related clinical signs and symptoms to 4 = severe clinical signs and symptoms of the disease.

SECONDARY OUTCOMES:
Time to the development of a recurrent FMF attack in patients with resolved "marker" attacks | from Day 7 to the development of a recurrent FMF attack, up to 16 weeks
  Criteria of a recurrent FMF attack development after resolution of "marker" attack include simultaneous development of clinical and laboratory signs of the attack:
  * PGA score ≥ 2 assuming mild, moderate or severe disease activity (i.e. clinical signs), AND
  * CRP level ≥ 30 mg/L (serological signs).
  PGA is a 5-point scale: from 0 = no disease-related clinical signs and symptoms to 4 = severe clinical signs and symptoms of the disease.
Proportion of subjects with Physician Global Assessment (PGA) score < 2 during the study | Up to 16 weeks
  PGA score < 2 during the treatment period with RPH-104 compared to placebo in FMF subjects with colchicine inefficacy or intolerance.
  PGA is a 5-point scale from 0 = no disease-related clinical signs and symptoms to 4 = severe clinical signs and symptoms of the disease.
Proportion of subjects with partial response to treatment | Up to 16 weeks
  Partial response defined as Resolution of "marker" attack by Visit 2 (Day 7) but with development of recurrent attacks up to Visit 10 (Day 112).
  Criteria of resolution of a "marker" FMF attack include simultaneous clinical and laboratory signs of the attack resolution:
  * Physician Global Assessment (PGA) score < 2 (i.e. minimum or complete lack of clinical signs and symptoms) AND
  * CRP level ≤ 10 mg/L OR CRP reduction by ≥ 70% compared to baseline defined at enrollment to treatment period (Visit 1).
  Criteria of a recurrent FMF attack development after resolution of "marker" attack include simultaneous development of clinical and laboratory signs of the attack:
  * PGA score ≥ 2 assuming mild, moderate or severe disease activity (i.e. clinical signs), AND
  * CRP level ≥ 30 mg/L (serological signs).
  PGA is a 5-point scale: from 0 = no disease-related clinical signs and symptoms to 4 = severe clinical signs and symptoms of the disease.
Proportion of subjects with serological remission | Up to 16 weeks
  Proportion of subjects with serological remission (CRP ≤ 10 mg/L) throughout the study.
Proportion of subjects with normalized Serum Amyloid A (SAA) level | Up to 16 weeks
  Proportion of subjects with normalized serum amyloid A level (SAA < 10 mg/L) throughout the study
Proportion of subjects escalated to RPH-104 160 mg q2w dose | Up to 16 weeks
  In patients whose treatment group has been unblinded because of a confirmed attack or no "marker" attack resolution: the patients from RPH-104 group and those switching from placebo and receiving RPH-104 at 80 mg dose will be escalated to RPH-104 160 mg q2w.
Proportion of subjects receiving additional symptomatic therapy with Nonsteroidal anti-inflammatory drugs (NSAIDs), paracetamol or glucocorticoids due to FMF | Up to 16 weeks
  Proportion of subjects receiving additional symptomatic therapy with NSAIDs, paracetamol or glucocorticoids due to FMF
Change in inflammation parameters vs. baseline (CRP) | From baseline (Day 0) up to 18 weeks
  Change in CRP levels vs. baseline (Day 0)
Change in inflammation parameters vs. baseline (SAA) | From baseline (Day 0) up to 18 weeks
  Change in SAA levels vs. baseline (Day 0)
PGA score change compared to baseline | From baseline (Day 0) up to 18 weeks
  PGA score change compared to baseline (Day 0) during the study. PGA is a 5-point scale from 0 = no disease-related clinical signs and symptoms to 4 = severe clinical signs and symptoms of the disease.
Changes in patients' quality of life during the treatment period with RPH-104 | From baseline (Day 0) up to 18 weeks
  Change in quality of life vs. baseline (Day 0) based on Medical Outcome Short Form (12) Health Survey (SF-)12® questionnaire throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (14):
- Armenia (2):
  - Center of Medical Genetics and Primary Health Care, Yerevan
  - Mikaelyan Institute Of Surgery CJSC, Yerevan
- Georgia (2):
  - Inova LLC, Tbilisi
  - The First Medical Center Ltd., Tbilisi
- Russia (5):
  - Federal State Autonomous Educational Institution of Higher Education I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University), Moscow
  - Multidisciplinary Scientific and Clinical Center named after S.P. Botkin, Moscow
  - Medical Technologies Ltd, Saint Petersburg
  - Saint-Petersburg Pasteur Institute, Saint Petersburg
  - Terafarm, Llc, Stavropol
- Turkey (Türkiye) (5):
  - Hacettepe University Faculty of Medicine, Ankara
  - Gazi University Faculty of Medicine, Ankara
  - Akdeniz University Faculty of Medicine, Antalya
  - Istanbul University Istanbul Faculty of Medicine, Istanbul
  - Istanbul University Cerrahpasa Faculty of Medicine, Istanbul